CLINICAL TRIAL: NCT01175954
Title: Phase IV Study of Cognitive and Behavioral Effects of Lacosamide as Adjunctive Therapy in Patients With Partial Epilepsy
Brief Title: Cognitive and Behavioral Effects of Lacosamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Evan Fertig (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Evan Fertig, Director, Northeast Regional Epilepsy Group
Organization: Northeast Regional Epilepsy Group (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEREG-002
Record Dates: First submitted 2010-07-09; First posted 2010-08-05 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Epilepsy
Keywords: Partial Epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide Open-Label (Experimental): Lacosamide will be titrated starting from visit 1 for 2 weeks (50mg bid) and maintained at 100mg bid for the rest of the study period.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Lacosamide will be titrated starting from visit 1 for 2 weeks (50mg bid) and maintained at 100mg bid for the rest of the study period. Dose Adjustments allowed up to 400 mg/day.
  Other Names: Vimpat
Drug: Lacosamide — Lacosamide will be titrated starting from visit 1 for 2 weeks (50mg bid) and maintained at 100mg bid for the rest of the study period.
  Other Names: Vimpat

SUMMARY:
Primary Objective:

Null hypothesis: A 24-week trial of adjunctive Lacosamide does not produce a decline in cognitive, mood or quality of life measures.

To determine the cognitive and behavioral side effects of lacosamide in patients with partial epilepsy and follow them for a period of 24 weeks using a neuropsychological test battery drawing on tests commonly used and designed to maximize sensitivity to drug effects.

Secondary Objectives:

To determine if any significant changes in cognitive, mood or quality of life measures are dependent upon changes in seizure severity, neurotoxicity, adverse events, or Lacosamide dosage.

DETAILED DESCRIPTION:
The investigators will examine a group of patients with partial epilepsy (chronic seizures arising from one particular part of the brain) whose seizures have not been controlled. If they consent to the study, they will be followed for 4 weeks to get a baseline seizure frequency. The patients will take a battery of tests assessing attention, memory, cognitive speed, and language, and fill out some inventories to assess their mood and quality of life. They will then receive a new anti-epileptic drug, lacosamide, to add to whatever epilepsy medications they are currently taking. They will be closely followed for 24 weeks with regular doctor's visits to monitor their physical health and seizure control, and will complete an inventory assessing the frequency and severity of their seizures. During that period of time, the other medication will remain unchanged. At the end of the 24-week period they will re-take the battery of cognitive tests and mood and quality of life inventories. The cognitive, mood, and quality of life variables will be analyzed to determine if they change for the better or worse after the course of lacosamide treatment. Any changes will also be analyzed with respect to seizure frequency and severity and to adverse events or side effects from the addition of the lacosamide, as well as to lacosamide dosage. The investigators chose this design since it closely represents what the investigators do in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible for enrollment into the trial

* Age range 18-70
* Able and willing to provide written informed consent to participate in the study in accordance with the ICH and GCP guidelines, and per the judgement of the investigator be able to cooperate fully with neuropsychological testing
* Native English speaker or balanced bilingual
* Diagnosis of refractory partial onset epilepsy
* Historical mean seizure frequency of >/= 1 seizure per month on average during 6 months prior to Visit 1.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

* History of drug/alcohol abuse
* Females who are pregnant or are on an unapproved method of contraception
* Psychiatric disorder (Diagnosis of Bipolar Disorder, Schizophrenia, psychotic disorder , Major Depression requiring hospitalization in the past 2 years, or other psychological or behavioral condition which in the judgement of the investigator should exclude the subject from the study.
* No active suicidal plan/intent or active suicidal thoughts in the last 6 months
* Current use of antidepressant, anxiolytic, or antipsychotic agents
* Presence of any progressive,demyelinating, or degenerative neurological condition
* Diagnosis of psychogenic non-epileptic seizure disorder
* Traumatic brain injury within 6 months of enrollment or TBI with suspected cognition/memory changes after TBI that has not stabilized 6 months prior to enrollment
* Prior history of cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in Cognitive test scores | 30 weeks
  Changes in the composite measure of the cognitive test scores and in the composite measure of the mood/Quality Of Life scores from baseline (visit 1) to scores recorded at termination (visit 4).

SECONDARY OUTCOMES:
Relationship of Cognitive test scores with Seizure severity ,A-B Neurotoxicity,Adverse Events and Lacosamide Dosage | 30 weeks
  The relationship of the cognitive and mood/Quality Of Life composite measures to seizure severity, A-B Neurotoxicity, Adverse Events, and Lacosamide dosage

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Lancman, MD, Principal Investigator — Northeast Regional Epilepsy Group
Locations (1):
- Northeast Regional Epilepsy Group, Hackensack, New Jersey, United States

REFERENCES:
- [Derived] Lancman ME, Fertig EJ, Trobliger RW, Perrine K, Myers L, Iyengar SS, Malik M. The effects of lacosamide on cognition, quality-of-life measures, and quality of life in patients with refractory partial epilepsy. Epilepsy Behav. 2016 Aug;61:27-33. doi: 10.1016/j.yebeh.2016.04.049. Epub 2016 Jun 14. PMID 27315132